CLINICAL TRIAL: NCT03942809
Title: Clinical Evaluation of the Revised iLTS-D2 in Effectivity and Practicability
Brief Title: Clinical Evaluation of the Revised iLTS-D2
Acronym: iLTS-D2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Principal investigator, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JohannesGU-iLT
Record Dates: First submitted 2019-04-22; First posted 2019-05-08 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Airway Management
Keywords: Airway Morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effectiveness (Experimental): Evaluate the Effectiveness in insertion success, insertion times, influence of respiratory, cardiac and cerebral circulation
  Interventions: Device: Effectiveness

INTERVENTIONS:
Device: Effectiveness — Effectiveness and Practicability in anesthetized patient under controlled conditions

SUMMARY:
A interventional, non-randomized, controlled study to evaluate the revised iLTS-D2 in anesthetized patients.

DETAILED DESCRIPTION:
The revised Intubation laryngeal tube - disposable (iLTS-D) is a refined laryngeal tube, which allows a secondary intubation over the inserted laryngeal tube. The present study should reveal the effectiveness and practicability in anesthetized patients in the operation room.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery patients under general Anesthesia

Exclusion Criteria:

* Age <18 years
* Existing pregnancy
* Lack of consent
* inability to consent
* emergency patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Insertion time LT | in 30 seconds
  Insertion of the laryngeal tube

SECONDARY OUTCOMES:
Insertion time ET | in 60 seconds
  Insertion of the endotracheal tube
Rate of successful Intubation attempts | through study completion, an average of 120 seconds
  successful insertion and tracheal intubation
hemodynamics MAP | through study completion, an average of 360 seconds
  changes in MAP (mmHg) during cuff insufflation of laryngeal tube
hemodynamics Freq | through study completion, an average of 360 seconds
  changes in heart frequency (bpm)
hemodynamics rO2 | through study completion, an average of 360 seconds
  changes in cerebral oxygenation (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University Medical Center Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No